CLINICAL TRIAL: NCT07057128
Title: Descriptors of Neuropathic Pain and Its Association With Central Sensitization in Subacromial Pain Syndrome
Brief Title: Neuropathic Characteristics of Subacromial Pain Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Aslı Gökgöz Azak, Assistant Doctor, Department of Physical Medicine and Rehabilitation, Izmir City Hospital, Izmir City Hospital
Other Study IDs: SAPS-NP
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Neuropathic Pain; Central Sensitization; Subacromial Pain Syndrome
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This single-center observational study aims to investigate neuropathic pain descriptors and their relationship with central sensitization in patients diagnosed with subacromial pain syndrome (SAPS) who have had shoulder pain for at least 3 months. A total of 82 participants aged 19 years or older will be recruited from the Physical Medicine and Rehabilitation outpatient clinic of Izmir City Hospital. After obtaining informed consent, participants will complete validated questionnaires assessing pain severity (VAS), neuropathic pain characteristics (painDETECT), central sensitization (Central Sensitization Inventory), and shoulder function (SPADI). Range of motion will be measured using a goniometer. No imaging or invasive procedures will be performed. Using the central sensitization scale and pain detect, the presence or absence of the 7 pain descriptors will be investigated in patients with subacromial pain syndrome with or without central sensitization and neuropathic pain pattern and it will be investigated whether the contribution of hyperalgesia, one of these pain descriptors, to neuropathic pain and central sensitization in patients with subacromial pain syndrome is greater than the contribution of other pain descriptors.The results of this study are expected to provide insight into pain mechanisms and guide clinical management in patients with SAPS.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of subacromial pain syndrome (SAPS)
2. Age ≥ 19 years
3. Shoulder pain lasting for at least 3 months
4. Shoulder pain intensity rated as 3 or higher on the Visual Analog Scale (VAS) in the past week
5. Positive findings on the following clinical tests:

Hawkins-Kennedy test Painful arc test Infraspinatus muscle strength test

Exclusion Criteria:

1. History of inflammatory disease involving the shoulder joint
2. History of neurological disorders
3. History of prior shoulder surgery
4. Positive drop arm test
5. Loss of passive range of motion in the shoulder joint
6. Presence of muscle strength loss
7. Structurally confirmed shoulder pathology based on imaging studies
8. Full-thickness tear of the rotator cuff muscles
9. Presence of neurodeficit in the upper extremity
10. Diagnosis of cancer or active infection
11. Use of medications for neuropathic pain within the past 3 months for any reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted with 82 patients aged 19 years and older who have been admitted to the PTR outpatient clinic of Izmir City Hospital with shoulder pain and diagnosed with subacromial pain syndrome and who have had shoulder pain for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hyperalgesia | At baseline (single assessment)
  Hyperalgesia is defined as an exaggerated pain response to a painful stimulus that is disproportionate to the intensity of the stimulus. It is one of the pain descriptors assessed in the painDETECT questionnaire, which evaluates neuropathic pain features.It is one of the 7 questions in the painDETECT scale that evaluates neuropathic pain and is scored on a 6-point Likert scale and receives a score between 0-5.

SECONDARY OUTCOMES:
Pain Intensity | At baseline
  Pain severity will be assessed using the Visual Analog Scale (VAS). VAS is a 10 cm horizontal line with endpoints labeled "no pain" (0) and "worst imaginable pain" (10). Patients will mark a point on the line that best represents their current level of shoulder pain.
Neuropathic Pain | At baseline
  Neuropathic pain features will be assessed using the painDETECT questionnaire, which consists of 9 items. Two items evaluate pain pattern and radiation, and seven items assess descriptors such as burning, tingling, mechanical allodynia, paroxysmal pain, thermal hyperalgesia, numbness, and pressure-induced pain (hyperalgesia). Each descriptor is rated on a 0-5 scale. The total score helps determine the likelihood of neuropathic pain.
Central Sensitization | At baseline
  Central sensitization will be evaluated using the Central Sensitization Inventory (CSI), which includes 25 items scored from 0 (never) to 4 (always). A score of 40 or more suggests a high probability of central sensitization (81% sensitivity, 75% specificity).
Function | At baseline
  It will be evaluated with the shoulder pain and disability index (SPADI-Shoulder Pain and Disability Index). SPADI is a questionnaire with a total of 13 questions developed to measure disability associated with shoulder pain. In the subgroup of the questionnaire assessing pain, the patient is asked to rate the severity of pain during different activities in the past week by giving a score between zero (no pain) and 10 (most severe pain). In the sub-group assessing disability, the patient is asked to rate how much difficulty he/she has had during different activities in the last week by giving a score between zero (no difficulty at all) and 10 (receiving assistance). A score of zero indicates maximum well-being and a score of 130 indicates maximum ill health. The validity and reliability of the Turkish version of SPADI has been demonstrated.
Range of Motion Measurement | At baseline
  Active and passive shoulder range of motion (ROM) will be measured using a goniometer. The movements evaluated include flexion, extension, abduction, adduction, internal and external rotation.

IPD SHARING:
Plan to Share IPD: Undecided